CLINICAL TRIAL: NCT05019404
Title: Functional Anterior Temporal Lobectomy Via Minicraniotomy as a Novel Surgical Therapy for Temporal Lobe Epilepsy: a Randomized, Controlled Trial
Brief Title: Minimally Invasive Surgical Epilepsy Trial for Temporal Lobe Epilepsy
Acronym: MISET-TLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF2021LSK-194
Record Dates: First submitted 2021-07-09; First posted 2021-08-24 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-11

CONDITIONS: Temporal Lobe Epilepsy; Open Surgery; Minimally Invasive Surgery
Keywords: Temporal lobe epilepsy; Anterior temporal lobectomy; Functional anterior temporal lobectomy; Randomized controlled trial; Minicraniotomy
MeSH Terms: conditions — Epilepsy, Temporal Lobe | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Intervention Model Description: a single-center, prospective, single-blinded, double-arm, randomized, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors are blinded to the treatment throughout the entire study. Blinding is maintained by having patients wear large hats during the interview to obscure skin incision and providing patients strict instruction not to reveal treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional anterior temporal lobectomy (FATL) (Experimental): FATL via minicraniotomy is a new surgical approach, consisting of amygdalohippocampectomy and the lateral temporal lobotomy.
  Interventions: Procedure: Functional anterior temporal lobectomy (FATL)
- Anterior temporal lobectomy (ATL) (Active Comparator): ATL via large frontotemporal craniotomy is a conventional surgical approach, consisting of amygdalohippocampectomy and en bloc resection of the lateral temporal lobe.
  Interventions: Procedure: Anterior temporal lobectomy (ATL)

INTERVENTIONS:
Procedure: Functional anterior temporal lobectomy (FATL) — Patients are placed in the supine position with the head contralaterally rotated 30°. The 3D model of incision and bone flap is printed prior to surgery by the slicer software based on the MRI data. Slightly curve incision with the length of about 6 cm in the temporal region is marked according to the 3D model. Temporal craniotomy via small bone window with the diameter of about 3 cm is performed. From the temporal pole along T1 about 5 cm posteriorly, temporal horn is opened by dissecting the middle temporal gyrus. The head of temporal horn is exposed. The amygdala is resected. Then, the parahippocampal gyrus and hippocampus are en bloc resected. The lateral temporal lobotomy is easy due to large view following the removal of mesial structures. The lateral posterior temporal lobotomy is no more than 5 cm from the temporal pole.
  Arms: Functional anterior temporal lobectomy (FATL)
Procedure: Anterior temporal lobectomy (ATL) — Patients are placed in the supine position with the head contralaterally rotated 30°. Large frontotemporal craniotomy is performed. Question mark-shaped incision with the length of 20- 25 cm in the frontotemporal region is marked. The size of the bone flap is approximately 5×7 cm for the exposure of lateral temporal lobe. ATL consists of en bloc resection of the anterior 5 cm of lateral temporal lobe, followed by the removal of mesial structures including the amygdala, parahippocampal gyrus, and hippocampus.
  Arms: Anterior temporal lobectomy (ATL)

SUMMARY:
Temporal lobe epilepsy (TLE) is a chronically neurological disease characterized by progressive seizures. TLE is the most frequent subtype of refractory focal epilepsy in adults. Epilepsy surgery has proven to be very efficient in TLE and superior to medical therapy in two randomized controlled trials. According to the previous experience, the investigators use functional anterior temporal lobectomy (FATL) via minicraniotomy for TLE. To date, this minimally invasive open surgery has been not reported. The investigators here present a protocol of a prospective trail which for the first time evaluates the outcomes of this new surgical therapy for TLE.

DETAILED DESCRIPTION:
Temporal lobe epilepsy (TLE) is a chronically neurological disease characterized by progressive seizures, followed by a latency period of several years after various injuries including febrile seizures, infection, trauma, tumors, and vascular malformation. Hippocampal sclerosis is the most common histopathological finding. The macroscopic changes of TLE with hippocampal sclerosis include the diminished size, sclerosis, and reduced metabolism in mesial temporal structures (amygdala, hippocampus, and parahippocampal gyrus). The microscopic changes include neuronal loss, gliosis, and axonal reorganization. As TLE progresses, most of patients become resistant to current antiepileptic drugs. Therefore, TLE is the most frequent subtype of refractory focal epilepsy in adults.

Epilepsy surgery has proven to be very efficient for TLE and superior to medical therapy in two randomized controlled trials. Patients with surgical therapy have high seizure-free rate with the range of 60% to 80 % while less than 5% with medical treatment. Anterior temporal lobectomy (ATL) is the most frequently used approach for TLE. For patients with TLE, Engel suggested referral to ATL should be strongly considered. The decision analysis showed that ATL increased life expectancy and quality- adjusted life expectancy in patients with TLE compared with medical management. Nevertheless, ATL is performed by large frontotemporal craniotomy. Although complication rates after temporal lobectomy have decreased dramatically over time, ATL creates a large cavity with temporal lobe resected, causing potential complications such as bleeding, brain shifts and subdural collections. With the advances in minimally invasive surgery, surgical techniques of ATL for TLE need to be continuously improved.

For this reason, the investigators modify the surgical approach. Functional anterior temporal lobectomy (FATL) via minicraniotomy is established. Recently, 25 patients with TLE undergoing FATL obtained satisfactory outcomes in our center (unpublished data). To date, this new open surgery for TLE has been not reported. The safety and efficacy of FATL need to be verified. Therefore, the investigators here present a protocol of the minimally invasive surgical epilepsy trial for TLE (MISET-TLE) which for the first time evaluates the outcomes of FATL as a new surgical approach for TLE.

ELIGIBILITY:
Inclusion Criteria:

1. male or female aged between 18 and 60 years;
2. drug- resistant temporal lobe epilepsy, remaining seizures after two or more tolerated and appropriately chosen antiepileptic drugs;
3. monthly or more seizures during the preceding year prior to trial;
4. the full- scale intelligence quotient (IQ) more than 70, understanding and completing the trial;
5. signing the informed consent;
6. good compliance, at least 12- month follow- up after surgery.

Exclusion Criteria:

1. tumor in temporal lobe;
2. extratemporal epilepsy and temporal plus epilepsy;
3. drug- responsive epilepsy, seizure freedom with current drugs in recent one year;
4. pseudoseizures;
5. seizures arising from bilateral temporal lobes;
6. significant comorbidities including progressive neurological disorders, active psychosis, and drug abuse;
7. a full- scale IQ lower than 70, unable to complete tests;
8. previous epilepsy surgery;
9. poor compliance and inadequate follow- up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-25 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Surgery duration | At the end of the surgery.
  Surgery duration in hours, the time from the beginning of incising the skin to the finish of suturing the skin.
Blood loss | At the end of the surgery.
  Blood loss in millilitres during the operation.
Skin incision | At the end of the surgery.
  Length of skin incision in centimetres
Bone flap | At the end of the surgery.
  Size of bone flap in square centimeter
Postoperative hospital stay | Up to 1 month after surgery.
  Postoperative hospital stay in days, the time from the first postoperative day to discharge date.
Complications | Up to 1 year after epilepsy surgery
  The incidence of postoperative complications

SECONDARY OUTCOMES:
Seizure outcomes classified by the International League Against Epilepsy (ILAE) | Up to 1 year after epilepsy surgery
  Seizure outcomes are classified by the International League Against Epilepsy (ILAE). Specific seizure classifications: class 1, seizure-free; class 2, only auras, no other seizures; class 3, 1-3 seizure days per year with or without auras; class 4, ≥4 seizure days per year and ≥50% reduction in baseline numbers of seizure days, with or without auras; class 5, <50% reduction and ≤100% increase in baseline numbers of seizure days, with or without auras; class 6, >100% increase in baseline numbers of seizure days, with or without auras.
  Proportion of each class is calculated.
Seizure outcomes classified by the Engel | Up to 1 year after epilepsy surgery
  Seizure outcomes are also classified by the Engel classification: class 1, free from disabling seizures; class 2, rare disabling seizures (almost seizure free); class 3, worthwhile improvement; class 4, no worthwhile improvement.
  Proportion of each class is calculated.
Quality of life assessed by the Quality of Life in Epilepsy Inventory- 89 | Up to 1 year after epilepsy surgery
  Quality of life is evaluated by the epilepsy- specific Quality of Life in Epilepsy Inventory- 89 (QOLIE- 89). QOLIE-89 is one of the special inventories applied mostly to assess QOL in research protocols, especially in long-term prospective clinical investigations. QOLIE- 89 has 89 items, range of scores, 0 to 100, with higher scores indicating better QOL.

OTHER OUTCOMES:
Intelligence assessed by the Wechsler Adult Intelligence Scale | Up to 1 year after epilepsy surgery
  Intelligence is assessed by the Wechsler Adult Intelligence Scale IV (WAIS-IV). WAIS-IV provides four major domains: perceptual reasoning, processing speed, verbal comprehension, working memory. The WAIS-IV also provides two overall summary scores including a Full-Scale IQ and a General Ability Index (GAI), where FSIQ is a measurement of performance across all subcategories, but the GAI is more resistant to issues that might arise from cognitive impairment, allowing for a more precise and truthful analysis. Higher score means better outcome. Intelligence is classified according to the total score : 1) extremely abnormal with more than 130 points; 2) Exceptional: 120-129 points; 3) Higher than usual: 110-119 points; 4) Normal: 90-109 points; 5) Lower than usual: 80-89 points; 6) Boundary: 70-79 points; 7) Mental Retardation: lower than 69 points.
Depression assessed by Beck's Depression Inventory | Up to 1 year after epilepsy surgery
  Beck's Depression Inventory (BDI) with 21 items, range of scores, 0 to 63. Higher score means a worse outcome.
Anxiety assessed by the State-Trait Anxiety Inventory | Up to 1 year after epilepsy surgery
  The State-Trait Anxiety Inventory (STAI) with 40 items, range of scores, 20 to 80. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhang, PhD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] O'Dell CM, Das A, Wallace G 4th, Ray SK, Banik NL. Understanding the basic mechanisms underlying seizures in mesial temporal lobe epilepsy and possible therapeutic targets: a review. J Neurosci Res. 2012 May;90(5):913-24. doi: 10.1002/jnr.22829. Epub 2012 Feb 8. PMID 22315182
- [Background] Falowski SM, Wallace D, Kanner A, Smith M, Rossi M, Balabanov A, Ouyang B, Byrne RW. Tailored temporal lobectomy for medically intractable epilepsy: evaluation of pathology and predictors of outcome. Neurosurgery. 2012 Sep;71(3):703-9; discussion 709. doi: 10.1227/NEU.0b013e318262161d. PMID 22668889
- [Background] Jones AL, Cascino GD. Evidence on Use of Neuroimaging for Surgical Treatment of Temporal Lobe Epilepsy: A Systematic Review. JAMA Neurol. 2016 Apr;73(4):464-70. doi: 10.1001/jamaneurol.2015.4996. PMID 26926529
- [Background] Wiebe S, Blume WT, Girvin JP, Eliasziw M; Effectiveness and Efficiency of Surgery for Temporal Lobe Epilepsy Study Group. A randomized, controlled trial of surgery for temporal-lobe epilepsy. N Engl J Med. 2001 Aug 2;345(5):311-8. doi: 10.1056/NEJM200108023450501. PMID 11484687
- [Background] Engel J Jr, McDermott MP, Wiebe S, Langfitt JT, Stern JM, Dewar S, Sperling MR, Gardiner I, Erba G, Fried I, Jacobs M, Vinters HV, Mintzer S, Kieburtz K; Early Randomized Surgical Epilepsy Trial (ERSET) Study Group. Early surgical therapy for drug-resistant temporal lobe epilepsy: a randomized trial. JAMA. 2012 Mar 7;307(9):922-30. doi: 10.1001/jama.2012.220. PMID 22396514
- [Background] Chang EF, Englot DJ, Vadera S. Minimally invasive surgical approaches for temporal lobe epilepsy. Epilepsy Behav. 2015 Jun;47:24-33. doi: 10.1016/j.yebeh.2015.04.033. Epub 2015 May 24. PMID 26017774
- [Background] Engel J Jr, Wiebe S, French J, Sperling M, Williamson P, Spencer D, Gumnit R, Zahn C, Westbrook E, Enos B. Practice parameter: temporal lobe and localized neocortical resections for epilepsy. Epilepsia. 2003 Jun;44(6):741-51. doi: 10.1046/j.1528-1157.2003.48202.x. PMID 12790886
- [Background] Choi H, Sell RL, Lenert L, Muennig P, Goodman RR, Gilliam FG, Wong JB. Epilepsy surgery for pharmacoresistant temporal lobe epilepsy: a decision analysis. JAMA. 2008 Dec 3;300(21):2497-505. doi: 10.1001/jama.2008.771. PMID 19050193
- [Background] Tebo CC, Evins AI, Christos PJ, Kwon J, Schwartz TH. Evolution of cranial epilepsy surgery complication rates: a 32-year systematic review and meta-analysis. J Neurosurg. 2014 Jun;120(6):1415-27. doi: 10.3171/2014.1.JNS131694. Epub 2014 Feb 21. PMID 24559222
- [Background] Wieser HG, Blume WT, Fish D, Goldensohn E, Hufnagel A, King D, Sperling MR, Luders H, Pedley TA; Commission on Neurosurgery of the International League Against Epilepsy (ILAE). ILAE Commission Report. Proposal for a new classification of outcome with respect to epileptic seizures following epilepsy surgery. Epilepsia. 2001 Feb;42(2):282-6. No abstract available. PMID 11240604
- [Background] Zhao Y, Ding C, Wang Y, Li Z, Zhou Y, Huang Y. Reliability and validity of a Chinese version of the Quality of Life in Epilepsy Inventory (QOLIE-89). Epilepsy Behav. 2007 Aug;11(1):53-9. doi: 10.1016/j.yebeh.2007.03.013. Epub 2007 May 10. PMID 17499025
- [Background] Brissart H, Planton M, Bilger M, Bulteau C, Forthoffer N, Guinet V, Hennion S, Kleitz C, Laguitton V, Mirabel H, Mosca C, Pecheux N, Pradier S, Samson S, Tramoni E, Voltzenlogel V, Denos M, Boutin M. French neuropsychological procedure consensus in epilepsy surgery. Epilepsy Behav. 2019 Nov;100(Pt A):106522. doi: 10.1016/j.yebeh.2019.106522. Epub 2019 Oct 15. PMID 31627076
- [Background] Schmeiser B, Wagner K, Schulze-Bonhage A, Mader I, Wendling AS, Steinhoff BJ, Prinz M, Scheiwe C, Weyerbrock A, Zentner J. Surgical Treatment of Mesiotemporal Lobe Epilepsy: Which Approach is Favorable? Neurosurgery. 2017 Dec 1;81(6):992-1004. doi: 10.1093/neuros/nyx138. PMID 28582572
- [Background] Tellez-Zenteno JF, Dhar R, Wiebe S. Long-term seizure outcomes following epilepsy surgery: a systematic review and meta-analysis. Brain. 2005 May;128(Pt 5):1188-98. doi: 10.1093/brain/awh449. Epub 2005 Mar 9. PMID 15758038
- [Background] Brotis AG, Giannis T, Kapsalaki E, Dardiotis E, Fountas KN. Complications after Anterior Temporal Lobectomy for Medically Intractable Epilepsy: A Systematic Review and Meta-Analysis. Stereotact Funct Neurosurg. 2019;97(2):69-82. doi: 10.1159/000500136. Epub 2019 Jul 9. PMID 31288240
- [Background] Bjellvi J, Flink R, Rydenhag B, Malmgren K. Complications of epilepsy surgery in Sweden 1996-2010: a prospective, population-based study. J Neurosurg. 2015 Mar;122(3):519-25. doi: 10.3171/2014.9.JNS132679. Epub 2014 Oct 31. PMID 25361484

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT05019404/Prot_SAP_000.pdf